CLINICAL TRIAL: NCT05203380
Title: Neuropsychologic Assessments of Dupilumab-Treated Adolescents With Moderate-to-Severe Atopic Dermatitis
Brief Title: Neuropsychologic Assessments of Dupilumab-Treated Adolescent Participants With Moderate-to-Severe Atopic Dermatitis
Acronym: NEURADAD
Status: Completed | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-AD-2024
Record Dates: First submitted 2022-01-05; First posted 2022-01-24 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Moderate-to-severe Atopic Dermatitis
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part A: Assessed in a single visit and no study-related treatment will be given.
- Part B: Patients in Part A may also enroll in Part B provided they meet the eligibility criteria.
  Interventions: Drug: dupilumab

INTERVENTIONS:
Drug: dupilumab — Weight based dosing for 16 weeks in accordance of United States prescribing information (USPI)
  Other Names: DUPIXENT®
  Groups: Part B

SUMMARY:
Primary Objective: Part A

* To quantify deficits in cognitive functioning in adolescents with moderate-to-severe AD, using the Conners' Continuous Performance Test 3rd Edition (CPT-3) d' T-score
* To determine the entry criterion (CPT-3 d' score) for Part B

Primary Objective: Part B

* To measure changes in cognitive functioning in adolescents with moderate-to-severe AD treated with dupilumab

Secondary Objectives

* To evaluate the relationship of cognitive and sensory functioning with severity of AD in adolescent AD patients
* To evaluate the relationship between changes in AD severity and changes in cognitive and sensory functioning scores following treatment with dupilumab (Part B only).

DETAILED DESCRIPTION:
Per protocol Study Stop Criteria, study has concluded with Part A. Part B was not initiated and no data were collected.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adolescent (12 - 17 years of age) Part A: at time of visit Part B: at time of screening visit
2. Diagnosis of atopic dermatitis (AD) according to American Academy of Dermatology consensus criteria; chronic AD Part A: first diagnosed at least 1 year prior to visit Part B: first diagnosed at least 1 year prior to the screening visit
3. EASI score ≥ 12 Part A: at time of visit Part B: at screening and baseline visits
4. IGA score ≥ 3 Part A: at time of visit Part B: at time of screening and baseline visits
5. Peak Pruritus NRS score ≥ 4 Part A: at time of visit Part B: at time of screening and baseline visits as defined in the protocol
6. The CPT-3 d' score for entry into Part B will be determined based on the distribution of the CPT-3 d' score from Part A
7. BSA of AD involvement ≥ 10% Part A: at time visit Part B: at screening and baseline visits
8. Part B Only: Documented recent history (within 6 months of the screening visit) of inadequate response (in the opinion of the investigator) to topical AD medication(s) or for whom topical AD medications are medically inadvisable as defined in the protocol
9. Part B Only: Patient's stable use of a prescription topical medication regimen for AD lesions for at least 2 weeks prior to baseline as defined in the protocol

Key Exclusion Criteria:

1. Prior use of dupilumab Part A: within 6 months of visit Part B: within 6 months of screening
2. Skin diseases that could confound AD assessment as defined in the protocol
3. Treatment with methylphenidate, dexmethylphenidate, serdexmethylphenidate, amphetamine, dextroamphetamine, lisdexamfetamine, guanfacine, atomoxetine, clonidine, or viloxazine within 8 weeks or within 5 half-lives, whichever is longer, at visit
4. History of clinician-diagnosed attention-deficit/hyperactivity disorder (ADHD), autism spectrum disorder, epilepsy, major depressive disorder, mania or bipolar disorder, or any Diagnostic and Statistical Manual-V (DSM-V) psychotic disorder, such as schizophrenia
5. Evidence of substance abuse, including alcohol and nicotine, in the past 2 years
6. Systemic antihistamine or nicotine use Part A: within the week prior to the visit Part B: during the week prior to screening
7. Part B Only: Active helminthic infections; suspected or high risk of helminthic infection, unless clinical and (if necessary) laboratory assessments have ruled out active infection before baseline
8. Part B Only: At baseline, presence of any conditions listed as criteria for study drug discontinuation
9. Part B Only: Treatment with high potency or super-potent TCS within 14 days prior to baseline

NOTE: Other protocol defined inclusion/exclusion criteria apply

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents with moderate-to-severe atopic dermatitis (AD) will be assessed for quantifying deficits in cognitive functioning at a single visit only and no study-related treatment will be offered.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Proportion of AD patients with a Conner's CPT-3 d' T-score ≥ 60 | Day 1
  Part A
  Conners' Continuous Performance Test-3 (CPT-3): an objective test of attention and impulsivity that has been validated in individuals aged 8 years and older. The primary efficacy outcome measure (d' T-score) is a measure of "signal detectability" with respect to inattentiveness, that is, the respondent's ability to differentiate non-targets (ie, the letter X) from targets (ie, all other letters), and is calculated as: d' = z-score ("False Alarm") - z-score ("Hit"). "T scores" refer to a distribution of the d' statistic such that the mean is 50 and the standard deviation (SD) is 10. Lower d' T-score values indicate worse performance.
Mean change from baseline in Conner's CPT-3 d' T-score | At week 16
  Part B
  Conner's CPT-3 d' T-scoring as stated above.

SECONDARY OUTCOMES:
Correlation of values for Conners' Continuous Performance Test 3rd Edition (CPT-3) scores (d' T-score, Commission Errors, Omission Errors, and Reaction Time) with AD disease severity based on Eczema Area and Severity Index (EASI) | Day 1
  Part A
  Conner's CPT-3 d' T-scoring as stated above.
  EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, apulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator or designee on a scale of 0" (absent) through "3" (severe). In addition, the area of AD involvement will be assessed as a percentage by body area of head, trunk, upper limbs, and lower limbs, and converted to a score of 0 to 6.
Correlation of values for Conners' CPT-3 scores with AD disease severity based on Body Surface Area (BSA) | Day 1
  Part A
  Conner's CPT-3 d' T-scoring as stated above.
  BSA affected by AD is assessed for each section of the body using the rule of nines (the possible highest score for each region is: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and will be reported as a percentage of all major body sections combined.
Correlation of values for Conners' CPT-3 scores with AD disease severity based on Peak Pruritus Numeric Rating Scale (NRS) | Day 1
  Part A
  Conner's CPT-3 d' T-scoring as stated above.
  Peak Pruritus NRS is a simple assessment tool that patients will use to report the average intensity of their pruritus (itch), both maximum and average intensity, during a 24-hour recall period; maximum itch intensity on a scale of 0 - 10 (0 = no itch; 10 = worst itch imaginable).
Correlation of values for Conners' CPT-3 scores with AD disease severity based on Skin Pain Numeric Rating Scale (SP-NRS) | Day 1
  Part A
  Conner's CPT-3 d' T-scoring as stated above.
  SP-NRS is a validated, self-administered PRO measuring the skin pain severity at its worst with a recall period of 24 hours pain severity in adults and adolescents. This single-item questionnaire uses an 11-point scale, which ranges from "0-No pain" to "10-Worst pain possible." Skin pain severity based on SP-NRS can be categorized as: clear (0), mild (1-3), moderate (5-6), severe (7-9), and very severe (10).
Correlation of values for Conners' CPT-3 scores with AD disease severity based on Patient-Reported Outcomes Measurement Information System Pediatric Sleep Disturbance Questionnaire (PROMIS Pediatric Sleep Disturbance) | Day 1
  Part A
  Conner's CPT-3 d' T-scoring as stated above.
  PROMIS sleep disturbance questionnaire is used to measure self-reported perceptions of sleep quality, sleep depth, and restoration. This includes perceived difficulties getting to sleep and staying asleep, as well as sleep satisfaction. Parent-reported sleep.
Correlation of values for Conners' CPT-3 scores with AD disease severity based on Children's Dermatology Life Quality Index (CDLQI) | Day 1
  Part A
  Conner's CPT-3 d' T-scoring as stated above.
  CDLQI is a validated questionnaire designed to measure the impact of skin disease on the quality of life (QoL) in children over a recall period of the past week. 9 of the 10 questions are scored by (0) Not answered/not at all, (1) only a little, (2) quite a lot to (3) very much. Question 7 has a possible response of (3) prevented school. The sum of the score of each question has a maximum of 30 and a minimum of 0. The higher the score the greater the impact on QoL. CDLQI can be a percentage of the maximum possible score of 30.
Correlation of values for Conners' CPT-3 scores with AD disease severity based on Hospital Anxiety and Depression Scale (HADS) | Day 1
  Part A
  Conner's CPT-3 d' T-scoring as stated above.
  HADS is an instrument for screening anxiety and depression in non-psychiatric populations; repeated administration also provides information about changes in a patient's emotional state. HADS consists of 14 items, 7 each for anxiety and depression symptoms; possible scores range from 0 to 21 for each subscale. The following cut-off scores are recommended for both subscales: 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression.
Correlation of values for Conners' CPT-3 scores with AD disease severity based on Investigator's Global Assessment (IGA) | Day 1
  Part A
  Conner's CPT-3 d' T-scoring as stated above.
  IGA is an instrument used for rapid and easy assessment of atopic dermatitis disease lesional severity globally based on a 5-point scale with range from 0-4, (0 = Clear, 1 = Almost clear, 2 = Mild disease, 3 = Moderate disease and 4 = Severe disease).
Correlation of values for Adult/Adolescent Sensory Profile (AASP) Sensory Sensitivity Score with AD disease severity based on EASI | Day 1
  Part A
  AASP is a 60-item self-report questionnaire measuring sensory responsiveness patterns in six different sensory modalities, including taste/smell, movement, visual, touch, activity and auditory processing. Patients complete the AASP by responding to each item with a five-point Likert scale (1 = almost never, 2 = seldom, 3 =occasionally, 4 = frequently, or 5 = always). Higher scores in each quadrant represented stronger preference to adopt certain types of sensory responsiveness patterns. The quadrant score can be categorized into one of the 5 categories, indicating how a particular patient's score compares to people in the same age group (adolescents of age 11-17 years) without disabilities: much less than most people, less than most people, similar to most people, more than most people, much more than most people.
  EASI measuring as stated above.
Correlation of values for AASP Sensory Sensitivity Score with AD disease severity based on BSA | Day 1
  Part A
  AASP scoring as stated above. BSA scoring as stated above.
Correlation of values for AASP Sensory Sensitivity Score with AD disease severity based on Peak Pruritus NRS | Day 1
  Part A
  AASP scoring as stated above. Peak Pruritus NRS scaling as stated above.
Correlation of values for AASP Sensory Sensitivity Score with AD disease severity based on SP-NRS | Day 1
  Part A
  AASP scoring as stated above. SP-NRS scaling as stated above.
Correlation of values for AASP Sensory Sensitivity Score with AD disease severity based on PROMIS Pediatric Sleep Disturbance Questionnaire | Day 1
  Part A
  AASP scoring as stated above. PROMIS Pediatric sleep disturbance scaling as stated above.
Correlation of values for AASP Sensory Sensitivity Score with AD disease severity based on CDLQI | Day 1
  Part A
  AASP scoring as stated above. CDLQI scoring as stated above.
Correlation of values for AASP Sensory Sensitivity Score with AD disease severity based on HADS | Day 1
  Part A
  AASP scoring as stated above. HADS scoring as stated above.
Correlation of values for AASP Sensory Sensitivity Score with AD disease severity based on IGA | Day 1
  Part A
  AASP scoring as stated above. IGA scoring as stated above.
Correlation of values for Stroop Interference Score with AD disease severity based on EASI | Day 1
  Part A
  Stroop Color and Word Test (SCWT) is a test used to measure selective inhibition, the ability to attend to certain environmental stimuli while inhibiting other stimuli. Stroop Interference scores are calculated from the number of correctly identified items in the three trials. Higher Stroop Interference scores represent poorer performance and suggests impaired executive functioning.
  EASI scoring as stated above.
Correlation of values for SCWT Interference Score with AD disease severity based on BSA | Day 1
  Part A
  SCWT scoring as stated above. BSA scoring as stated above.
Correlation of values for Stroop Interference Score with AD disease severity based on Peak Pruritus NRS | Day 1
  PART A
  SCWT scoring as stated above. Peak Pruritus NRS scoring as stated above.
Correlation of values for Stroop Interference Score with AD disease severity based on SP-NRS | Day 1
  Part A
  SCWT scoring as stated above. SP-NRS scoring as stated above.
Correlation of values for Stroop Interference Score with AD disease severity based on PROMIS Pediatric Sleep Disturbance Questionnaire | Day 1
  Part A
  SCWT scoring as stated above. PROMIS scoring as stated above.
Correlation of values for Stroop Interference Score with AD disease severity based on CDLQI | Day 1
  Part A
  SCWT scoring as stated above. CDLQI scoring as stated above.
Correlation of values for Stroop Interference Score with AD disease severity based on HADS | Day 1
  Part A
  SCWT scoring as stated above. HADS scoring as stated above.
Correlation of values for Stroop Interference Score with AD disease severity based on IGA | Day 1
  Part A
  SCWT scoring as stated above. IGA scoring as stated above.
Determine the appropriate minimal Conners' CPT-3 d-prime T score | Day 1
  Used as an entrance criterion into Part B
Correlation of change in AD disease severity based on EASI with change in Conners' CPT-3 score | Up to Week 16
  Part B
  EASI scoring as stated above. Conners' CPT-3 scoring as stated above.
Correlation of change in AD disease severity based on BSA with change in Conners' CPT-3 score | Up to Week 16
  Part B
  BSA scoring as stated above. Conners' CPT-3 scoring as stated above.
Correlation of change in AD disease severity based on Peak Pruritus NRS with change in Conners' CPT-3 score | Up to Week 16
  Part B
  Peak Pruritus NRS scoring as stated above. Conners' CPT-3 scroring as stated above.
Correlation of change in AD disease severity based on SP-NRS with change in Conners' CPT-3 score | Up to Week 16
  Part B
  SP-NRS scoring as stated above. Conners' CPT-3 scoring as stated above.
Correlation of change in AD disease severity based on PROMIS Pediatric Sleep Disturbance with change in Conners' CPT-3 score | Up to Week 16
  Part B
  PROMIS scoring as stated above. Conners' CPT-3 scoring as stated above.
Correlation of change in AD disease severity based on CDLQI with change in Conners' CPT-3 score | Up to Week 16
  Part B
  CDLQI scoring as stated above. Conners' CPT-3 scoring as stated above.
Correlation of change in AD disease severity based on HADS with change in Conners' CPT-3 score | Up to Week 16
  Part B
  HADS scoring as stated above. Conners' CPT-3 scoring as stated above.
Correlation of change in AD disease severity based on IGA with change in Conners' CPT-3 score | Up to Week 16
  Part B
  IGA scoring as stated above. Conners' CPT-3 scoring as stated above.
Correlation of change in AD disease severity based on EASI with AASP Sensory Sensitivity Summary Score | Up to Week 16
  Part B
  EASI scoring as stated above. AASP scoring as stated above.
Correlation of change in AD disease severity based on BSA with AASP Sensory Sensitivity Summary Score | Up to Week 16
  Part B
  BSA scoring as stated above. AASP scoring as stated above.
Correlation of change in AD disease severity based on Peak Pruritus NRS with AASP Sensory Sensitivity Summary Score | Up to Week 16
  Part B
  Peak Pruritus NRS scoring as stated above. AASP scoring as stated above.
Correlation of change in AD disease severity based on SP-NRS with AASP Sensory Sensitivity Summary Score | Up to Week 16
  Part B
  SP-NRS scoring as stated above. AASP scoring as stated above.
Correlation of change in AD disease severity based on PROMIS Pediatric Sleep Disturbance with AASP Sensory Sensitivity Summary Score | Up to Week 16
  Part B
  PROMIS scoring as stated above. AASP scoring as stated above.
Correlation of change in AD disease severity based on CDLQI with AASP Sensory Sensitivity Summary Score | Up to Week 16
  Part B
  CDLQI scoring as stated above. AASP scoring as stated above.
Correlation of change in AD disease severity based on HADS with AASP Sensory Sensitivity Summary Score | Up to Week 16
  Part B
  HADS scoring as stated above. AASP scoring as stated above.
Correlation of change in AD disease severity based on IGA with AASP Sensory Sensitivity Summary Score | Up to Week 16
  Part B
  IGA scoring as stated above. AASP scoring as stated above.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (10):
- United States (10):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Arizona Allergy & Immunology Research, Gilbert, Arizona
  - Pediatric Skin Research, LLC, Coral Gables, Florida
  - Skin Research of South Florida, LLC, Miami, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - DermAssociates, LLC, Rockville, Maryland
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

REFERENCES:
- [Derived] Paller AS, Gonzalez ME, Barnum S, Jaeger J, Shao L, Ozturk ZE, Korotzer A. Attentiveness and mental health in adolescents with moderate-to-severe atopic dermatitis without ADHD. Arch Dermatol Res. 2024 Jul 30;316(8):497. doi: 10.1007/s00403-024-03210-x. PMID 39080094